CLINICAL TRIAL: NCT03023943
Title: The Effects of Instrument Assisted Soft Tissue Mobilization on Proprioception
Brief Title: The Effects of IASTM and Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Weiqing Ge, Associate Professor, Youngstown State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 072-2017
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IASTM group (Experimental): Intervention will be 10 minutes of GT1 instrument application at anterior thigh using sweep technique.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization — Intervention will be 10 minutes of GT1 instrument application at anterior thigh using sweep technique.
  Other Names: IASTM

SUMMARY:
The research design will be single group pretest-posttest design. The subject will be instructed to position the knee joint to a position previously set by the experimenter. Intervention will be 10 minutes of GT1 instrument application at anterior thigh using sweep technique.

ELIGIBILITY:
Inclusion Criteria:

* male or female, age 18 to 65.

Exclusion Criteria:

* sensory impairments or a present contraindications to IASTM which include cancer, burn scars, kidney dysfunction, pregnancy, varicose veins, osteoporosis, body art, chronic regional pain syndrome, polyneuropathies, fractures, autoimmune disorders, diabetes, vitamin C & D/Calcium deficiencies, rheumatoid arthritis, ankylosing spondylitis, congestive heart failure, acute inflammation, lymphedema, flu or illness with flu-like symptoms, and medications (anticoagulant, steroids, hormone replacements, NSAIDS, fluoroquinolone antibiotics, herbal supplements).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Proprioception determined using the reposition error | 5 minutes
  Proprioception will be determined by measuring the reposition error of the knee joint. The subject will be instructed to position the knee joint to a position (flexion) previously set by the experimenter at 30 degree flexion. The difference will be calculated as the reposition error. The position of the knee joint will be measure using a goniometer. An alternative is to use an App (e.g. Angle Meter) on a smart phone or an iPad for accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hripko, Study Director — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States